CLINICAL TRIAL: NCT01130129
Title: The Effects of Plant Bioactives on Platelet Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Quadram Institute Bioscience (Other)
Collaborators: European Union (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IFR02/2009
Record Dates: First submitted 2010-05-24; First posted 2010-05-25 (Estimated); Last update posted 2013-03-06 (Estimated); Status verified 2013-03

CONDITIONS: Healthy
Keywords: Flavonoids; Platelets
MeSH Terms: interventions — Flavonoids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ex-vivo treatment of platelets (Experimental): Ex-vivo treatment of platelets
  Interventions: Other: Ex-vivo treatments with flavonoids

INTERVENTIONS:
Other: Ex-vivo treatments with flavonoids — Ex-vivo treatment of platelets with a range of flavonoids

SUMMARY:
Consumption of a diet rich in fruit and vegetables is associated with a reduced risk of cardiovascular disease and the protective effect may be due to polyphenolic compounds contained within these foods. The mechanism by which polyphenols exert this effect is not clearly understood but research has focused on their potential to affect platelet function. The purpose of this study is to quantify the anti-clotting activity of a range of plant food extracts and component compounds.

DETAILED DESCRIPTION:
A single sample of whole blood will be collected from 15 male or female volunteers aged between 18 and 65 years. After collection whole blood will be treated with a range of flavonoids to evaluate their effects on platelet function.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Aged 18 - 65 years.
* BMI > 19.5 and < 35
* Non-smokers

Exclusion Criteria:

* Pregnancy or have been pregnant within the last 12 months
* Parallel participation in another research project which involves dietary intervention
* Participation in another research project which has involved blood sampling within the last four months unless the total amount of combined blood from both studies does not exceed 470 mls.
* Has donated or intends to donate blood within 16 weeks prior to during the Study period.
* Depressed or elevated blood pressure measurements (<90/50 or 95/50 if symptomatic or >160/100)
* Any person related to or living with any member of the study team
* Diabetics
* Taking regular prescribed and/or non-prescribed medication (excluding oral contraceptive and HRT).
* Known bleeding disorders.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Identification of flavonoids that exert a significant anti-clotting effect | within 4hours

CONTACTS AND LOCATIONS:
Overall Officials: Paul Kroon, phD, Principal Investigator — Quadram Institute Bioscience
Locations (1):
- Institute of Food Research, Norwich, Norfolk, United Kingdom